CLINICAL TRIAL: NCT02567552
Title: Randomized Clinical Trial Comparing Endometrial Transformation With Subcutaneous Progesterone (Prolutex) 25 mg/Day Versus Intramuscular Progesterone (Prontogest) 50 mg/Day
Brief Title: Clinical Trial Comparing Endometrial Transformation With Subcutaneous Progesterone Versus Intramuscular Progesterone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IVI Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1412-BCN-087-AB; 2015-000290-12 (EudraCT Number)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-02

CONDITIONS: Reproductive Techniques, Assisted
Keywords: endometrial receptivity; endometrial predecidualization; endometrial genomics; endometrial receptivity array
MeSH Terms: conditions — Helping Behavior

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Masked samples for histological evaluation and assessment of gene expression
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolutex (Experimental): Subcutaneous progesterone
  Interventions: Drug: Subcutaneous progesterone
- Prontogest (Active Comparator): Intramuscular progesterone
  Interventions: Drug: Intramuscular progesterone

INTERVENTIONS:
Drug: Subcutaneous progesterone — subcutaneous progesterone 25 mg/day
  Other Names: Prolutex
  Arms: Prolutex
Drug: Intramuscular progesterone — intramuscular progesterone 50 mg/day
  Other Names: Prontogest
  Arms: Prontogest

SUMMARY:
Study the endometrial predecidualization by using subcutaneous progesterone 25 mg/day versus intramuscular progesterone 50 mg/day, to determine whether there are differences in the endometrial transformation and endometrial receptivity.

DETAILED DESCRIPTION:
The aim of this study is to compare predecidualization and endometrial receptivity as gene expression by using subcutaneous progesterone 25 mg/day versus intramuscular progesterone 50 mg/day in healthy women of childbearing age. Both, the two drugs and the doses administered in this clinical trial, are routine clinical practice.

A controlled ovarian stimulation will be previously performed and following routine clinical practice for 10-12 days at standard doses of subcutaneous FSH 150-225 IU/day, according to BMI and number of antral follicles. A GnRH antagonist shall be administered, being initiated according to donor's follicular growth from greater or equal14 mm diameter follicles. Final maturation shall be performed with a bolus of GnRH agonist when there exist at least 3 follicles greater or equal17 mm diameter, and therefore performing follicular puncture 36 hours after the bolus of agonist has been administered.

If the donor meets the inclusion criteria, she will be informed of the study and, if she agrees, she will sign the informed consent. Randomization shall be performed in 2 arms; arm 1 will be administered subcutaneous progesterone 25 mg/day (Prolutex; Angelini, Spain), and arm 2, intramuscular progesterone 50 mg/day (Prontogest IBSA, Italy). In each arm 12 donors (ITT population) will be included.

The randomization to a treatment group shall be performed the day the follicular puncture has been programmed. To that purpose, a randomized consecutive sampling will be used by means of assignment tables. The medication will be administered by a person not involved in the assessments and responsible for group assignment, data centralization and drug assignment.

At day 5 (5 days after follicular puncture):endometrial thickness measurement by means of transvaginal ultrasound and perform endometrial biopsy and take two samples: 1 sample to Anatomical Pathology and 1 sample to Endometrial Receptivity Array (ERA).

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 18 and 34 years
* BMI between 18 and 28 kg/m2
* Endometrial thickness > 7 mm the day of progesterone treatment initiation (day of follicular puncture)
* Follicular maturation with a single bolus of GnRH agonist
* Egg donors who undergo a cycle of ovarian stimulation in the IVI Barcelona Centre
* Egg donors selected in accordance with the requirements of Law 14/2006 of 26 May 2006 on Assisted Human Reproduction Techniques
* Informed consent has been signed and dated

Exclusion Criteria:

* Known allergy to progesterone formulations or their excipients
* Known allergy to estrogens
* Known thrombophilias
* Alcohol, drug or psychotropic medication dependence
* Concurrent participation in another study
* Concomitant medication that may interfere with the study medication and ovarian stimulation
* Failure to comply with the requirements for egg donors in accordance with Law 14/2006 of 26 May 2006 on Assisted Human Reproduction Techniques

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustín B Boluda, Principal Investigator — IVI Barcelona
Locations (1):
- IVI Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prolutex | Prontogest
Started | 12 | 12
Completed | 12 | 11 (dropout by pain in the puncture site)
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolutex | Prontogest | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.92 (5.32) | 25.58 (2.39) | 26.25 (4.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 21.76 (2.88) | 23.12 (2.79) | 22.44 (2.86)
Height [Mean (Standard Deviation); unit: cm] | 166.75 (5.10) | 162.08 (3.50) | 164.42 (4.90)
Weight [Mean (Standard Deviation); unit: Kg] | 61.00 (10.05) | 61.00 (8.55) | 61.00 (9.12)
Blood Progesterone Level [Mean (Standard Deviation); unit: ng/ml] — Blood progesterone level in Day -2
  ng/ml | 1.31 (0.85) | 1.44 (0.77) | 1.37 (0.79)
Blood Estradiol Level [Mean (Standard Deviation); unit: pg/ml] — Blood Estradiol Level in day -2
  pg/ml | 2020.35 (998.36) | 2464.33 (1144.19) | 2262.52 (1078.94)
Blood LH level [Mean (Standard Deviation); unit: pg/ml] — Blood LH level in day -2
  pg/ml | 1.25 (0.45) | 1.24 (0.91) | 1.25 (0.70)
Endometrial Thickness [Mean (Standard Deviation); unit: mm] — Endometrial Thickness in day 0
  mm | 8.88 (1.98) | 9.58 (1.61) | 9.23 (1.80)

OUTCOME MEASURES:

1. Primary Outcome: Predecidual Transformation
Description: Histologic dating of the endometrium at day 5: early secretory phase, media secretory phase or late secretory phase
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 11
participants
  early secretory phase | 1 | 2
  media secretory phase | 7 | 8
  late secretory phase | 4 | 1
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; Test type: Other; p = 0.3395, Chi-squared

2. Primary Outcome: Decidualization of Stromal Cell
Description: Rate of transformation of endometrial stromal fibroblasts into specialized secretory decidual cells (three categories: less than 25%, between 26% and 50%, and over 50%)
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 11
participants
  <25% of stromal cell | 3 | 2
  25-50% of stromal cell | 3 | 7
  > 50% of stromal cell | 6 | 2
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; Test type: Other; p = 0.1523, Chi-squared

3. Primary Outcome: Endometrial Maturation Using Noyes' Criteria
Description: Endometrial dating of luteal phase days according to the Noyes criteria
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 11
days | 9.08 (2.23) | 7.64 (2.01)
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; comparison between groups; Test type: Other; p = 0.1189, t-test, 2 sided

4. Primary Outcome: Endometrial Gene Expression
Description: Gene expression profile of endometrial
Time Frame: 5 days
Population: We assessed the gene expression of 238 endometrial genes to detect differences in gene expression between treatments.
  This analysis could not be performed in 1 patient of the prolutex group because of the poor quality of the sample collected
Measure: Number; unit: Endometrial genes
Units Other Than Participants: Endometrial genes
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 11 | 11
Number analyzed (Endometrial genes) | 238 | 238
Endometrial genes
  differential expressed genes | 28 | 28
  the same trend of gene expression | 210 | 210

5. Secondary Outcome: Endometrial Thickness
Description: Endometrial thickness measurement by means of transvaginal ultrasound.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 12
mm | 8.46 (2.66) | 9.61 (1.24)
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; Test type: Other; p = 0.2042, t-test, 2 sided

6. Secondary Outcome: Blood Estradiol Level
Description: Blood estradiol level on the day of follicular puncture
Time Frame: day 0
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 11
pg/mL | 1384.06 (1122.80) | 1208.58 (502.96)
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; Test type: Other; p = 0.6262, t-test, 2 sided

7. Secondary Outcome: Blood Progesterone Level
Description: Blood progesterone level on the day of follicular puncture
Time Frame: day 0
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 12
ng/mL | 14.40 (6.63) | 10.92 (6.88)
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; Test type: Other; p = 0.2301, t-test, 2 sided

8. Secondary Outcome: Blood LH Level
Description: Blood Luteinizing hormone level on the day of follicular puncture
Time Frame: day 0
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 12
pg/mL | 2.32 (0.89) | 2.75 (2.08)
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; Test type: Other; p = 0.5118, t-test, 2 sided

9. Secondary Outcome: Blood Estradiol Level
Description: Blood estradiol level 5 days after progesterone treatment
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 11
pg/mL | 257.88 (150.65) | 246.45 (106.90)
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; Test type: Other; p = 0.8371, t-test, 2 sided

10. Secondary Outcome: Blood Progesterone Level
Description: Blood progesterone level 5 days after progesterone treatment
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 11
ng/mL | 3.16 (1.00) | 11.04 (5.21)
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; Test type: Other; p < 0.0001, t-test, 2 sided

11. Secondary Outcome: Blood LH Level
Description: Blood Luteinizing hormone level 5 days after progesterone treatment
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 11
pg/mL | 1.30 (0.60) | 2.92 (5.36)
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; Test type: Other; p = 0.3107, t-test, 2 sided

12. Secondary Outcome: Number of Participants With Side Effects During the Study
Description: Number of Participants with side effects during the study"
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 12 | 12
participants | 5 | 4
Statistical Analysis 1: Comparison: Prolutex vs Prontogest; Test type: Other; p = 0.5, Fisher Exact

13. Primary Outcome: Endometrial Gene Expression Difference
Description: Genes with a significantly high gene expression difference (adj-p-value < 0.05, Fold Change>3)
Time Frame: 5 days
Population: We assessed the expressed genes with a significantly high gene expression difference between treatments (adj-p-value < 0.05, Fold Change>3) This analysis could not be performed in 1 patient of the prolutex group because of the poor quality of the sample collected
Measure: Number; unit: Endometrial genes
Units Other Than Participants: Endometrial genes
Arm/Group | Prolutex | Prontogest
Number analyzed (Participants) | 11 | 11
Number analyzed (Endometrial genes) | 238 | 238
Endometrial genes
  expressed genes with fold change > 3 | 4 | 4
  expressed genes without or with fold change < 3 | 234 | 234

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Prolutex | Prontogest
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolutex (N=12) | Prontogest (N=12)
Pain in injection site (General disorders) | 0 (0) | 4 (6) — Pain in injection site
Discomfort in injection site (General disorders) | 3 (6) | 0 (0) — Discomfort in injection site
Breast inflammation (Reproductive system and breast disorders) | 2 (2) | 0 (0) — Breast inflammation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes